CLINICAL TRIAL: NCT04312139
Title: Development of a Serum and Cellular Biomarkers Cluster for the Assessment of Degenerative Aortic Valve Stenosis Progression.
Brief Title: Serum and Cellular Biomarkers for Aortic Valve Stenosis
Acronym: AthenaValve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Naval Hospital of Athens (Unknown); Biomedical Research Foundation of the Academy of Athens (Unknown); University of Oxford (Other)
Responsible Party: Principal Investigator, Konstantinos Toutouzas, Professor of Cardiology, National and Kapodistrian University of Athens
Other Study IDs: Τ2ΕΔΚ-01683
Record Dates: First submitted 2020-03-14; First posted 2020-03-18 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Calcific Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve, Calcification of
Keywords: aortic valve stenosis; calcific aortic valve disease; aortic stenosis; biomineralization; calcification; cardiovascular calcification; serum diagnostics; multiplex ELISA; LC-MS/MS; bioinformatics; disease progression; Integrated proteomics-metabolomics-transcriptomics; Mass cytometry; Flow cytometry; Immune cells
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve, Calcification of; Calcinosis; Disease Progression | interventions — Echocardiography; Liquid Chromatography-Mass Spectrometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum from peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Fast progressors of Aortic Valve Stenosis: 50 patients that retrospectively demonstrated fast progression from moderate to severe aortic valve stenosis: echocardiographic dVmax>0.25 m/sec/year (difference in transaortic Vmax).
  Interventions: Other: Untargeted LC/MS and LC-MS/MS
- Slow progressors of Aortic Valve Stenosis: 50 patients that retrospectively demonstrated slow progression from moderate to severe aortic valve stenosis: echocardiographic dVmax<0.15 m/sec/year (difference in transaortic Vmax).
  Interventions: Other: Untargeted LC/MS and LC-MS/MS
- Prospective Moderate Aortic Valve Stenosis: 100 consecutive prospectively enrolled patients with moderate aortic valve stenosis. Plus 20 patients accounting for 20% drop-out rate, total prospective cohort = 120 patients.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Computerized Tomography Aortic Valve Calcium Score; Other: Targeted LC/MS and LC-MS/MS; Diagnostic Test: multiplex ELISA
- Negative calcium score group: 50 patients at intermediate to high risk for Cardiovascular Disease (CVD) and negative aortic valve and coronary calcium score at CT scan, prospectively followed-up. Plus 10 patients accounting for 20% drop-out rate, total control cohort = 60 patients.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Computerized Tomography Aortic Valve Calcium Score; Other: Targeted LC/MS and LC-MS/MS; Diagnostic Test: multiplex ELISA

INTERVENTIONS:
Diagnostic Test: Echocardiography — Baseline and prospective follow-up echocardiography
  Groups: Negative calcium score group; Prospective Moderate Aortic Valve Stenosis
Diagnostic Test: Computerized Tomography Aortic Valve Calcium Score — Baseline and prospective follow-up CT calcium score of aortic valve
  Groups: Negative calcium score group; Prospective Moderate Aortic Valve Stenosis
Other: Untargeted LC/MS and LC-MS/MS — Serum samples untargeted proteomics and metabolomics
  Groups: Fast progressors of Aortic Valve Stenosis; Slow progressors of Aortic Valve Stenosis
Other: Targeted LC/MS and LC-MS/MS — Serum samples targeted proteomics and metabolomics
  Groups: Negative calcium score group; Prospective Moderate Aortic Valve Stenosis
Diagnostic Test: multiplex ELISA — Implementation of novel multiplex ELISA assay on serum samples of aortic valve stenosis prospective cohort.
  Groups: Negative calcium score group; Prospective Moderate Aortic Valve Stenosis

SUMMARY:
AthenaValve aims to develop and initial validate a novel serum diagnostic kit, for the assessment of severity and prognosis of progression of aortic valve stenosis (AS, a devastating disease without early diagnosis and medical treatment). Two independent clinical cohorts of patients will provide serum samples, along with tissue and serum of a validated animal model of the disease for evaluation of the early stages, in order to develop and validate a multiplexed Enzyme-linked Immunosorbent Assay kit (multiplex ELISA). Advanced bioinformatics analysis will facilitate the selection of the most promising molecules from integrated proteomics-transcriptomics-metabolomics data. The novel biomarkers will help clinicians to early diagnose patients at high risk and will pave the way for the experimental implementation of promising pharmaceutical therapies.

Moreover, AthenaValve aims to shed light on the systemic cellular interplay of the same patients, by analyzing the circulating immune cell phenotypes of the subgroups of rapid and slow progression patients

DETAILED DESCRIPTION:
The deposition of calcium salts in the arterial wall and the heart valves is a commonly occurring phenomenon associated with increasing age and various pathological factors. A particular case is the calcification of the aortic valve, which is accompanied by gradual stenosis leading to heart failure. As a result, causes significant morbidity and a dramatic increase in mortality if not treated surgically or via transcatheter intervention. It affects approximately 2% of the population over the age of 65, being the third cause of death in this population. It numbers about 100 surgeries per 100,000 person-years in the decade and 180000 patients each year are candidates for percutaneous aortic valve implantation (TAVI) in the US, Canada, and European Union.

Characteristic of the disease is that it remains even today without a diagnosis at the critical early stages and all existing therapies have failed to slow or reverse the damage when applied in the final stages. Previous experimental studies suggested that existing drugs may be more effective if given early in the disease course. At the time when the aortic stenosis becomes evident on echocardiography or Computerized Tomography (CT), underlying biochemical and molecular lesions have already developed. Moreover, among the aortic valve stenosis patients, it is unknown who will rapidly evolve to a dynamic narrowing of the valve and previous research studies report significantly diverse progression rates among patients, with approximately 20-25% demonstrating more than double rates. Thus, the Achilles heel of the therapeutic management of patients is the lack of early diagnosis and disease progression prognosis.

Under a combination of pathological effects by factors such as hypertension, diabetes mellitus and dyslipidemia in patients with a possible genetic predisposition, impairment of the normal structure and function of endothelium occurs, which progressively leads to the disease of the underlying valve tissue. Local acidosis and accumulation of oxidative oxygen radicals cause damage to membrane phospholipids, oxidation of cholesterol and proteins, which lose their normal quaternary structure and degrade. The gradual deposition of phosphate and calcium carbonate salts over the pathological proteins leads to calcification of the valve tissue. Intense inflammatory reaction with activation of bone marrow and infiltration of tissue with immunocompetent cells accompanies the damage: macrophages, B and T lymphocytes, mast cells infiltrate and actively contribute to the disease. Within this environment, inflammatory cytokines secreted from the inflammatory cells lead to activation of embryonic cell pathways that help to further enhance the calcification through the conversion of resident fibroblasts to active osteoblasts, which actively deposit calcium salts through extracellular vesicles.

In the disease, multiple cell types and distant organs are involved (liver - cholesterol metabolism, spleen and bone marrow - immune response activation) and the damage is expected to release fragments of biological and biochemical substances in the blood circulation. Hence, the disease is expected to be reflected in changes in serum protein. It is possible to detect proteins and metabolites in the blood serum in appropriately selected patients, prospectively enrolled and monitored through the course of aortic valve stenosis. An optimal subgroup description of patients with rapid or slow disease progression can reveal important information for future clinical diagnostic and prognostic use. Moreover, the disease is characterized by cellular infiltration of a plethora of known and unknown immune cells that contribute to the disease. Thus, the discovery of novel cellular phenotypes linked to disease progression can help delineate important clinical aspects.

The purposes of Athena Valve are:

(A) Collection of data on the progression of calcification and aortic valve stenosis, description of subpopulations with rapid and slow progression and record of clinical events.

(B) The bioinformatics analysis of data from combined transcriptomics-metabolomics-proteomics of diseased animal model aortic valve tissue in the early, intermediate and final stages, in comparison with existing patient multi-omics databases, in order to investigate candidate molecules - "drivers" of the damage with a causal relationship.

(C) The differential proteomic analysis of patient sera samples with severe aortic valve stenosis, retrospectively defined as rapid versus slow disease progressors and control group of individuals without aortic valve stenosis and severe calcification.

(D) The differential metabolomic analysis of patient sera samples with severe aortic valve stenosis, retrospectively defined as rapid versus slow disease progressors and control group of individuals without aortic valve stenosis and severe calcification.

(E) To obtain the differential profile of circulating immune cells among patients.

(F) The integrated bioinformatics data analysis of differential patient serum proteome and metabolome enriched with the results of the animal model and existing databases from other patients, to determine the most probable - causally related molecules with disease progression in a molecular network.

(G) Utilization of the more important protein targets for the development of a novel detection assay for multiple protein targets in blood serum by multiplex ELISA based on the results of the bioinformatics analysis.

(H) Application of the new assay multiplex ELISA in paired serum samples of patients with moderate to severe aortic stenosis and control group of individuals without aortic valve stenosis and severe calcification, prospectively enrolled and monitored, initial validation of the assay and review of its diagnostic performance.

Brief Methodology:

Two independent clinical cohorts will provide necessary data and serum samples. The first, a retrospective cohort of patients with severe aortic valve stenosis will define serum, echocardiographic and clinical differences among subgroups with different progression rates. The second cohort, prospectively developed, will confirm the retrospectively obtained clinical and echocardiographic data and provide baseline and follow-up measurements of aortic valve calcification (CT calcium score). Paired baseline and follow-up serum samples will validate serum targets from the retrospective cohort. Patients will be assessed with echocardiography annually and with follow-up CT at 2 and 5 years from enrollment.

Retrospective proteomics will be done with untargeted Liquid Chromatography/Mass Spectrometry (LC/MS) and metabolomics with untargeted Liquid Chromatography-tandem Mass Spectrometry (LC-MS/MS) in Serial Reaction Monitoring (SRM) mode. Prospective proteomics and metabolomics will be quantitative and targeted. Blood samples will be immediately frozen and stored to -80 C.

Moreover, peripheral blood mononuclear cells will be isolated and cryopreserved at -80 C with differential density centrifugation. Cell populations will be analyzed utilizing mass cytometry, flow cytometry, cell sorting, and molecular methods.

For pathophysiological enrichment, a modified New Zealand rabbit model for aortic stenosis will be used in a longitudinal protocol of tissue harvesting in the early, intermediate and late-stage disease (corresponding to inflammation - calcification and subsequent valve stenosis).

ELIGIBILITY:
Inclusion Criteria:

* Retrospective cohort: patients with severe aortic valve stenosis in echocardiography:

  • Vmax > 4 m/sec and mean Gradient >40 mmHg and/or Aortic Valve Area indexed (AVAi) < 0.6 cm2/m2 and/or Velocity index <0.25 whichever worse, with available complete past echocardiographic follow-up (>2 past studies) indicating disease progression, by the same performing physician.
* Prospective cohort: patients with moderate aortic valve stenosis in echocardiography:

  * Vmax 3-4 m/sec and mean Gradient 25-40 mmHg and/or AVAi 0.6-0.9 cm2/m2,
  * Where inconsistent: Velocity index = 0.25-0.50.
  * Technical details: Optimal doppler measurements obtained by the best feasible echocardiographic window (demonstrating at least 2 windows, where possible including right parasternal with or without pencil probe).
* Prospective Control group: patients at intermediate to high risk for CVD according to atherosclerotic risk factors assessment - Heart Score

Exclusion Criteria:

* Echocardiographic Stroke Volume indexed (SVi) <35 ml/m2
* Bicuspid aortic valve
* Stenosis of rheumatic etiology
* More than mild aortic valve regurgitation
* More than mild mitral valve regurgitation
* More than mild mitral stenosis
* Severe pulmonary hypertension
* Chronic ischemic heart failure with Ejection Fraction < 45%
* Right heart failure (based on the echocardiographic assessment of Right Ventricle Dimension, Tricuspid Annular Plane Systolic Excursion, tricuspid annular velocity, and clinical syndrome)
* Acutely decompensated Heart Failure with preserved Ejection Fraction <4 weeks
* N-terminal-pro hormone Brain Natriuretic Peptide (NT-proBNP)> 900 pg/ml for ages 60-75, NT-pro-BNP > 1800 pg/ml for ages >75 years
* Presence of chronic systematic inflammatory disease
* Presence of autoimmune disease
* Active malignancy
* History of chemotherapy past 3 years
* Any history of thoracic radiotherapy
* Active treatment with monoclonal antibodies
* Under-treated hypertension
* Under-treated metabolic or endocrine disease
* Acute infection (<4 weeks)
* Any acute inflammation (<4 weeks)
* Unstable angina - myocardial infarction past 3 moths
* Stage 4 or 5 Chronic Kidney Disease (as defined by CKD-EPI derived estimated Glomerular Filtration Rate or 24hr urine measurement)
* Any acute renal failure <4 weeks
* Stroke past 3 months
* Any disabling stroke
* Surgery except for minor procedures past 3 months
* Poor mobility/immobilization
* Life expectancy < 3 years for any reason
* Difficulty in following follow-up protocol for any reason

For the control group:

* Known coronary artery disease
* Any heart valve disease, excluding minor valve regurgitation
* Any heart failure
* Pulmonary Hypertension
* Peripheral artery disease
* Presence of chronic systematic inflammatory disease
* Presence of autoimmune disease
* Active malignancy
* History of chemotherapy past 3 years
* Any history of thoracic radiotherapy
* Active treatment with monoclonal antibodies
* Under-treated hypertension
* Under-treated metabolic or endocrine disease
* Acute infection (<4 weeks)
* Any acute inflammation (<4 weeks)
* Stage 4 or 5 Chronic Kidney Disease, as defined by the Chronic Kidney Disease - Epidemiology Collaboration (CKD-EPI) derived estimated Glomerular Filtration Rate or 24hr urine measurement
* Any acute renal failure <4 weeks
* Any stroke
* Surgery except for minor procedures past 3 months
* Poor mobility/immobilization
* Life expectancy < 3 years for any reason
* Difficulty in following follow-up protocol for any reason

Ages: 60 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with moderate and severe tricuspid aortic valve stenosis of degenerative etiology.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
multiplex ELISA kit Sensitivity | 5 years
  Overall multiplex ELISA kit sensitivity for the detection of fast aortic valve stenosis progression (dVmax>0.25 m/sec/year)
multiplex ELISA kit Specificity | 5 years
  Overall multiplex ELISA kit specificity for the detection of fast aortic valve stenosis progression (dVmax>0.25 m/sec/year)

SECONDARY OUTCOMES:
Fast progressors percentage | 5 years
  Percentage of patients with echocardiographic aortic valve stenosis fast progression (dVmax>0.25 m/sec/year)
Severe AS percentage | 5 years
  Percentage of patients having echocardiographic Aortic Valve Area < 0.6 cm2/m2
Coronary Artery Disease progression percentage | 5 years
  Percentage of angiographically significant stable Coronary Artery Disease (CAD) treated with percutaneous coronary intervention or coronary artery bypass grafting, in patients without previous CAD.
Major Adverse Cardiovascular Events rate | 5 years
  Composite Major Adverse Cardiovascular Events (MACE), percentage of patients with cardiac death or non-fatal myocardial infarction or non-fatal stroke.

OTHER OUTCOMES:
Differential PBMC profile | 5 years
  ROC curve of circulating cell subpopulations discriminating patients from healthy volunteers and fast from slow progressors

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos P Toutouzas, Professor, Principal Investigator — First Department of Cardiology, Athens Medical School, NKUA
Locations (2):
- Greece (2):
  - First Department of Cardiology, University of Athens, Medical School. Hippocratio Hospital, Athens, Attica
  - Naval Hospital of Athens, Athens